CLINICAL TRIAL: NCT07144592
Title: The Effects of a Solution-Focused Approach on Psychosocial Adjustment and Treatment Compliance in Individuals Diagnosed With Schizophrenia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Principal Investigator, Fatih Sahin, doctor, Muş Alparslan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 167678
Record Dates: First submitted 2025-08-06; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: SCHIZOPHRENIA 1 (Disorder); Psychosocial Adaptation; Treatment Adherence
Keywords: treatment adherence; Schizophrenia; solution-focused therapy,; psychiatric nursing
MeSH Terms: conditions — Treatment Adherence and Compliance; Schizophrenia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Solution-Focused Approach Program) (Experimental): A 6-week solution-focused approach program will be applied to the experimental group.
  Interventions: Behavioral: solution-oriented approach program
- control group (No Intervention: Usual Care at Community Mental Health Center) (No Intervention): No intervention will be applied to the control group

INTERVENTIONS:
Behavioral: solution-oriented approach program — The solution-focused nursing intervention applied to the experimental group in the study was planned as individual sessions, consisting of one session per week, lasting a total of six weeks. The interventions were based on the principles of solution-focused brief therapy, focusing on the individual's strengths, past coping experiences, and current resources. The interviews aimed to identify exceptions, build positive future expectations, set small but achievable goals, strengthen hope, and increase the individual's ability to utilize their internal resources. Each session used structured open-ended questions, scaling techniques, and future-oriented solution scenarios to support the individual's psychosocial adjustment and motivation for treatment.
  Arms: experimental group (Solution-Focused Approach Program)

SUMMARY:
The aim of this study is to evaluate the effects of a solution-focused approach-based individual intervention on psychosocial adjustment and treatment adherence in individuals diagnosed with schizophrenia.

The study will be conducted as a randomized controlled trial including 60 clinically stable individuals diagnosed with schizophrenia according to DSM-5 criteria and registered at a Community Mental Health Center affiliated with a university hospital. Participants will be randomly assigned to an experimental group (n=30) and a control group (n=30).

The experimental group will receive one individual solution-focused therapy session per week for six weeks. The control group will receive usual care only. Data will be collected using a Personal Information Form, the Psychosocial Adjustment Scale (PSSAS), and the Medication Adherence Scale (MARS).

DETAILED DESCRIPTION:
Objective:

Schizophrenia is a chronic psychiatric disorder that significantly affects thought, emotion, and behavior, often limiting social functioning, treatment adherence, and integration into daily life. There is an increasing need for person-centered, empowering, and brief intervention models in psychiatric nursing. This study aims to determine the effects of a solution-focused approach (SFA)-based individual intervention on psychosocial adjustment and treatment adherence in individuals with schizophrenia.

Study Design:

This research will use a pretest-posttest randomized controlled experimental design with a control group.

Study Population:

The study will include 60 individuals diagnosed with schizophrenia according to DSM-5 diagnostic criteria, considered clinically stable, and registered at a Community Mental Health Center affiliated with a university hospital in Türkiye. Participants will be randomly assigned to an experimental group (n=30) or a control group (n=30) using computer-assisted randomization.

Intervention:

Experimental Group: Participants will receive individual solution-focused therapy sessions once per week for six consecutive weeks. The sessions will emphasize individual strengths, recall positive coping experiences, support future goal setting, and provide guidance on repeating effective solutions.

Control Group: Participants will receive no additional intervention beyond usual care.

Outcome Measures:

Data will be collected with the following instruments:

Personal Information Form

Psychosocial Adjustment Scale (PSSAS)

Medication Adherence Scale (MARS)

Statistical Analyses:

Planned analyses will include independent samples t-tests, paired t-tests, and ANCOVA.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with schizophrenia according to DSM-5 diagnostic criteria,

Being between 18 and 65 years of age,

Being literate and verbally communicative,

Being clinically stable (not exhibiting symptoms of acute psychosis),

Being registered with a Community Mental Health Center (CMHC) and receiving regular services,

Being cognitively competent enough to participate in individual interviews during the research process,

Being an individual currently receiving psychiatric treatment and taking medication,

Agreeing to participate voluntarily in the study and signing a written informed consent form.

Exclusion Criteria:

* those who do not meet the inclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-10-25 (Estimated)

PRIMARY OUTCOMES:
pretest (6-week solution-focused approach before the intervention) | Baseline (1 week before intervention)]
  1. Psychosocial Adjustment (PSSAS)
  Description: Measured with the Psychosocial Adjustment Scale (PSSAS), which assesses social relationships, daily life management, and coping with stress. Scores range from 0 to 180; higher scores indicate better psychosocial adjustment.
  Time Frame: Baseline (within 1 week before intervention)
  Unit of Measure: Total score (0-180)
pretest (6-week solution-focused approach before the intervention) | Baseline (within 1 week before intervention)
  2. Medication Adherence (MARS)
  Description: Measured with the Medication Adherence Scale (MARS), which assesses adherence to prescribed pharmacological treatment. Scores range from 0 to 10; higher scores indicate better medication adherence.
  Time Frame: Baseline (within 1 week before intervention)
  Unit of Measure: Total score (0-10)

SECONDARY OUTCOMES:
posttest (After the 6-week solution-focused approach intervention) | 6 weeks after baseline (post-intervention)
  1. Psychosocial Adjustment Post-Intervention (PSSAS)
  Description: Psychosocial Adjustment Scale (PSSAS). Scores range from 0 to 180; higher scores indicate better psychosocial adjustment.
  Time Frame: 6 weeks after baseline (post-intervention)
  Unit of Measure: Total score (0-180)
posttest (After the 6-week solution-focused approach intervention) | Post-intervention (6 weeks after completion of the intervention)
  2. Medication Adherence Post-Intervention (MARS)
  Description: Medication Adherence Scale (MARS). Scores range from 0 to 10; higher scores indicate better medication adherence.
  Time Frame: Post-intervention (6 weeks after completion of the intervention)
  Unit of Measure: Total score (0-10)

CONTACTS AND LOCATIONS:
Locations (1):
- Community Mental Health Center, Muş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
will be shared at the end of the research